CLINICAL TRIAL: NCT00212862
Title: Dosing and Outcomes Study of Erythropoietic Stimulating Therapies
Brief Title: Dosing and Outcomes Study of Erythropoietic Stimulating Therapies in Patients With Chemotherapy Induced Anemia
Acronym: DOSE
Status: Completed | Type: Observational
Sponsor: Ortho Biotech Products, L.P. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004561; ABT-OP-03-02 (Other: Ortho Biotech Products, L.P.)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Anemia; Cancer
Keywords: Anemia; Cancer; Epoetin alfa; Darbepoetin alfa; Registry
MeSH Terms: conditions — Anemia; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chemotherapy induced anemia
  Interventions: Other: Patients with chemotherapy induced anemia

INTERVENTIONS:
Other: Patients with chemotherapy induced anemia — Physicians are instructed to continue to treat all patients according to their own best clinical judgment, but to submit information on the parameters and outcomes of this treatment to the database. Patients will have to fill the questionaire at the time of enrollment and baseline.

SUMMARY:
The purpose of this study is to describe patient characteristics, treatment patterns, and clinical outcomes in adult patients with cancer who are receiving erythropoiesis-stimulating therapy (EST).

DETAILED DESCRIPTION:
The Dosing and Outcomes Study of Erythropoietic Stimulating Therapies (DOSE) is a prospective, observational multicenter registry of approximately 1200 adult cancer patients receiving treatment with EST; eg, epoetin alfa or darbepoetin alfa. The planned duration of the DOSE Registry is three years. Based on initial results, the registry sponsor may elect to extend the duration of the registry.This study does not specify treatment protocols, require any particular assignment of patients to treatment protocols, or in any other way require participating physicians to alter their practice patterns. Participating physicians are instructed to continue to treat all patients according to their own best clinical judgment, but to submit information on baseline patient characteristics, treatment patterns, and clinical outcomes. Baseline determinations will include patient demographics, tumor and treatment type, hematologic parameters, and patient reported outcomes. Data will be collected over the 16-week study period with regard to EST treatment, hematologic outcomes and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer who are being treated with an erythropoiesis-stimulating therapy (EST) for anemia of cancer or cancer-related treatment
* Must be EST ''naive'' globally or must have been off treatment with an EST for at least 90 days
* Must speak and read english and be able to answer the type of simple questions presented in the patient questionnaires
* If the patient is identified for the study while an inpatient, they must be able to be followed for up to 16 weeks
* The patient must give consent to participate in the registry by signing the informed consent form

Exclusion Criteria:

* Patients currently participating in any other clinical study of EST (however, the patient may be undergoing treatment under an investigational cancer treatment protocol)
* Have or had been on dialysis for end stage renal disease in the past
* Has myelodysplasia or any myelodysplastic syndrome
* Patients are known to need stem cell transplant
* Patient who will self-administer the epoetin alfa or darbepoetin alfa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being treated with an erythropoiesis-stimulating therapy for chemotherapy induced anemia.
Sampling Method: Non-Probability Sample
Enrollment: 2130 (Actual)
Dates: Start 2003-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To document patient characteristics and patterns of clinical management | Up to 3 years
  The clinical management includes changes in chemotherapy, radiation, bleeding, missed EST doses.

SECONDARY OUTCOMES:
To assess the relationships between patient characteristics, treatment patterns and outcomes | Up to 3 years
To measure economic impacts, and quality of life | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- [Result] Larholt K, Pashos CL, Wang Q, Bookhart B, McKenzie RS, Piech CT. Dosing and Outcomes Study of Erythropoiesis-Stimulating Therapies (DOSE) : a registry for characterizing anaemia management and outcomes in oncology patients. Clin Drug Investig. 2008;28(3):159-67. doi: 10.2165/00044011-200828030-00003. PMID 18266401